CLINICAL TRIAL: NCT05803785
Title: A Phase 1, Open Label, Ascending Dose Study to Evaluate the Safety of BBC1501 Administered by Intravitreal Injection for Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Safety of BBC1501 Intravitreal Injection in Patients With Neovascular Age-Related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Benobio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBRP11001-101
Record Dates: First submitted 2023-03-12; First posted 2023-04-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BBC1501 1.25ug (Experimental): Cohort 1; open-label, non-randomized, single administration
  Interventions: Drug: BBC1501
- BBC1501 2.5ug (Experimental): Cohort 2; open-label, non-randomized, single administration
  Interventions: Drug: BBC1501
- BBC1501 5ug (Experimental): Cohort 3; open-label, non-randomized, single administration
  Interventions: Drug: BBC1501

INTERVENTIONS:
Drug: BBC1501 — BBC1501 solution for Intravitreal injection

SUMMARY:
This open-label study is being conducted to evaluate the initial safety and tolerability of BBC1501 IVT in patients with nAMD. The primary objective of this study is to evaluate the safety and tolerability of 3 ascending doses of IVT BBC1501 in patients with nAMD. The secondary objective of this study is to exploratory of BBC1501 efficacy following 3 ascending dose of BBC1501 in nAMD patient.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to provide voluntary written informed consent on the approved ICF, understand the study requirements, and are willing to follow and complete all the study required procedures.
* Male or female aged ≥ 50 years.
* Participants who as per investigator's judgements are non-responders to at least 2 prior anti-VEGF treatment for nAMD in the study eye
* Active CNV lesions, secondary to nAMD as confirmed with SD-OCT (or SS-OCT), FFA and fundus photography (FP) in the study eye.
* Best corrected visual acuity (BCVA) between 60 and 21 letters, inclusive, in the study eye using ETDRS testing or BCVA between 20/60 and 20/400 letters, inclusive, in the study eye by Snellen chart
* Participant has CST of at least 300 uM with presence of intraretinal and/or subretinal fluid
* Participants who have had a washout period of at least six weeks prior to first administration of the IMP for any IVT anti-VEGF medication and, who in the opinion of the investigator, have disease sufficiently stable to enable this interval.

Key Exclusion Criteria:

* Use of any of the following treatments or anticipated use of any of the following treatments to the study eye:
* Intravitreal or periocular corticosteroid, within 90 days prior to Visit 1 (Day 1) and throughout the study.
* Glaucoma, evidenced by an IOP of > 21 mmHg, or chronic hypotony (< 6 mmHg) in the study eye.
* Evidence of any other ocular disease other than nAMD in the study eye that may confound the outcome of the study (eg, active diabetic retinopathy, posterior uveitis, pseudovitelliform macular degeneration, moderate/severe myopia).
* Participants with advanced nAMD and no prognosis of BCVA as per Investigator's judgement (e.g. due to macular OCT signs of atrophy or photoreceptors disruption, or macular/foveal subretinal hemorrhage).
* Need for ocular surgery in the study eye during the course of the study.
* YAG laser capsulotomy within 30 days prior to Visit 1 (Day 1) in the study eye.
* Intraocular surgery, including lens removal or laser, within 90 days prior to Visit 1 (Day 1) in the study eye.
* Ocular or periocular infection in either eye.
* Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye.
* Media opacity that would limit clinical visualization, intravenous fluorescein angiography, or spectral-domain optical coherence tomography (SD-OCT) evaluation in the study eye.
* History of herpetic infection in the study eye or adnexa.
* Presence of known active toxoplasmosis, inactive toxoplasmosis or toxoplasmosis scar in either eye.
* Presence of any form of ocular malignancy including choroidal melanoma in either eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of ophthalmic and systemic TEAEs, during study period | Every week up to 4 weeks
  To evaluate the safety and tolerability of a single IVT dose of BBC1501 at 4 weeks after dose.To characterize ocular and non-ocular safety by the incidence of treatment-emergent adverse events (AEs) (new or worsening from baseline) summarized categorically by system organ class and/or preferred term.
Assessment of ophthalmic and systemic TEAEs, during study period | every 4 weeks up to 12 weeks
  To evaluate the safety and tolerability of a single IVT dose of BBC1501 at 12 weeks after dose.To characterize ocular and non-ocular safety by the incidence of treatment-emergent adverse events (AEs) (new or worsening from baseline) summarized categorically by system organ class and/or preferred term.

SECONDARY OUTCOMES:
Mean change in Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA from baseline | Baseline, Week4
  Assessment ETDRS change from baseline by Optical Coherence Tomography(OCT)
Mean change in Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA from baseline | Baseline, Week12
  Assessment ETDRS change from baseline by Optical Coherence Tomography(OCT)
Number of patients who initiation of rescue therapy during study | Week1, Week12
  Exploratory using rescue therapy during study and follow-up period

OTHER OUTCOMES:
Change in CNV size according to fluorescein angiogram | Baseline, Week4
  Assessment CNV size change from baseline by Fundus fluorescein angiography(FFA)
Change in CNV size according to fluorescein angiogram | Baseline, Week12
  Assessment CNV size change from baseline by Fundus fluorescein angiography(FFA)
Changes in intra-or sub-retinal fluid measured as mean change in central retinal thickness or macula volume | Baseline, Week4
  Assessment Central retinal thickness from baseline by Spectral Domain Optical Coherence Tomography (SD-OCT)
Changes in intra-or sub-retinal fluid measured as mean change in central retinal thickness or macula volume | Baseline, Week12
  Assessment Central retinal thickness from baseline by Spectral Domain Optical Coherence Tomography (SD-OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Inhyun Lee, ph.D, Study Chair — Benobio Co., Ltd.
Locations (2):
- Australia (2):
  - Benobio Investigational site, Sydney, New South Wales
  - Sydney Hospital, Sydney

IPD SHARING:
Plan to Share IPD: No